CLINICAL TRIAL: NCT00418353
Title: Antenatal Betamethasone Compared to Dexamethasone - "BETACODE TRIAL"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Stony Brook University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20024615
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Respiratory Distress Syndrome; Intraventricular Hemorrhage; Neonatal Mortality
Keywords: Antenatal corticosteroids; Betamethasone; Dexamethasone; Premature
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — Dexamethasone

INTERVENTIONS:
Drug: Betamethasone(Celestone soluspan) and Dexamethasone

SUMMARY:
Antenatal corticosteroids result in substantial decrease in neonatal morbidity and mortality by specifically reducing the risk of respiratory distress syndrome, intraventricular hemorrhage and neonatal death among premature infants. No human randomized study has formally compared betamethasone and dexamethasone, the preferred corticosteroids for antenatal therapy, with regards to their effectiveness in reducing neonatal morbidities and mortality. Our objective was to compare betamethasone with dexamethasone in terms of effectiveness in reducing perinatal morbidities and mortality among preterm infants.

DETAILED DESCRIPTION:
We conducted a double blind placebo-controlled randomized trial of antenatal betamethasone compared to dexamethasone among women at risk of preterm deliveries at Stony Brook University Hospital from August 1, 2002 through July 31, 2004. We excluded women with clinical chorioamnionitis, major fetal structural anomalies, fetal chromosomal abnormalities, prior antenatal steroid exposure, and use of betamethasone or dexamethasone for other medical indications, quadruplets and higher order multiple gestation and those who declined enrollment. Consenting women were randomly allocated to one of two groups by the Pharmacy using computer generated random numbers. The statistical analysis was performed in accordance of the intention-to-treat principle. Student t test, Chi square and Fisher exact test were used for analysis. A P value of < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women in preterm labor with intact membranes
* Women with preterm premature rupture of membranes
* Women been delivered for fetal and maternal indications
* Gestational age between 24 and 33 6/7 weeks'.

Exclusion Criteria:

* Clinical chorioamnionitis
* known major fetal structural anomalies,
* known fetal chromosomal abnormalities,
* prior antenatal steroid exposure,
* quadruplets and higher order multiple gestation
* Women who declined enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2002-08; Study Completion 2005-04

PRIMARY OUTCOMES:
Respiratory distress syndrome
Intraventricular hemorrhage
Neonatal mortality

SECONDARY OUTCOMES:
Periventricular leukomalacia
Necrotizing enterocolitis
Neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Elimian, M.D, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Elimian A, Garry D, Figueroa R, Spitzer A, Wiencek V, Quirk JG. Antenatal betamethasone compared with dexamethasone (betacode trial): a randomized controlled trial. Obstet Gynecol. 2007 Jul;110(1):26-30. doi: 10.1097/01.AOG.0000268281.36788.81. PMID 17601892